CLINICAL TRIAL: NCT06392945
Title: Effects of Rhythmic Auditory Cueing Augments Cognitive Treadmill Walking Training on Community Walking Capacity, Walking Automaticity, and Social Participation in Individuals With Chronic Stroke: a Randomized Controlled Trial
Brief Title: Effects of Rhythmic Auditory Cueing Augments Cognitive Treadmill Walking Training in Individuals With Chronic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Li-Ling Chuang, Associated Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSTC 112-2314B-182-021
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: stroke; gait rehabilitation; rhythmic auditory cueing; cognitive training; treadmill
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Treadmill Walking Training with Rhythmic Auditory Cueing (CTW+RAC) group (Experimental): The CTW+RAC group will undertake progressive treadmill walking speed while performing a cognitive task with rhythmic auditory cueing (i.e., 110% of baseline cadence).
  Interventions: Device: Cognitive Treadmill Walking Training with Rhythmic Auditory Cueing (CTW+RAC) group
- Cognitive Treadmill Walking Training (CTW) (Active Comparator): The CTW group will receive cognitive training while walking at a progressive speed on the treadmill.
  Interventions: Device: Cognitive Treadmill Walking Training (CTW) group
- Treadmill Walking Training (TW) (Active Comparator): The TW group will train only in treadmill walking with progressive speed adjusted weekly.
  Interventions: Device: Treadmill Walking Training (TW)

INTERVENTIONS:
Device: Cognitive Treadmill Walking Training with Rhythmic Auditory Cueing (CTW+RAC) group — Participants in the CTW+RAC group participate in 12-session programs administered for 30 minutes each session, 3 times per week for 4 weeks. To increase adaptability to rhythmic auditory cueing prior to cognitive treadmill walking training, participants are required to keep stepping on their feet while listening to the auditory cueing using a metronome program (Metronome APP) for 5 minutes of warm up. Then they start walking on a treadmill with a target speed and perform a cognitive task concurrently while listening rhythmic auditory cueing. According to previous research, the target treadmill speed at week 1, week 2, week 3, and week 4 is gradually increased from 90%, 100%, 110%, to 120% baseline walking speed of comfortable walking on the ground. The beat of rhythmic auditory cueing using the Metronome APP on the smartphone is set at 110% of baseline cadence of comfortable walking on the ground based on a previous study in individuals with stroke.
  Arms: Cognitive Treadmill Walking Training with Rhythmic Auditory Cueing (CTW+RAC) group
Device: Cognitive Treadmill Walking Training (CTW) group — Participants in the CTW group will participate in 12-session programs administered for 30 minutes each session, 3 times per week for 4 weeks. They will start stepping on the ground at comfortable pace for 5 minutes of warm up. Then they will start walking on a treadmill with a target speed and perform a cognitive task concurrently without rhythmic auditory cueing. Same cognitive training and target treadmill speed will be used as the CTW+RAC group during cognitive dual-task treadmill walking. Three cognitive training programs will be the verbal fluency, arithmetic, and visual distinguish tasks. The target treadmill speed will be gradually increased from 90% at week 1, to 100% at week 2, to 110% at week 3, to 120% baseline walking speed of comfortable walking on the 10 meters walk test at week 4.
  Arms: Cognitive Treadmill Walking Training (CTW)
Device: Treadmill Walking Training (TW) — Participants in the TW group will participate in 12-session programs administered for 30 minutes each session, 3 times per week for 4 weeks. They will start stepping on the ground at comfortable pace for 5 minutes of warm up. Then they will start walking on a treadmill with a target speed only, without concurrent performing a cognitive task and no listening rhythmic auditory cueing. Same target treadmill speed will be used as the other two groups during treadmill walking. The target treadmill speed will be gradually increased from 90% at week 1, to 100% at week 2, to 110% at week 3, to 120% baseline walking speed of comfortable walking on the ground.
  Arms: Treadmill Walking Training (TW)

SUMMARY:
The first objective of this study is to examine the superiority of the combined rhythmic auditory cueing with cognitive treadmill training (combined group) in people with stroke as compared with the cognitive treadmill walking training (cognitive group) or treadmill walking training alone (treadmill group) (Aim 1). The study's second aim is to investigate the factors affecting the improvement in community walking capacity after interventions and to explore whether changes in community walking capacity are associated with changes in participation after interventions (Aim 2).

DETAILED DESCRIPTION:
A single-blind, randomized controlled trial is conducted at medical centers. Ninety stroke patients will be randomized to one of the three groups. All groups will receive interventions 30 minutes per time, 3 times a week, for 4 weeks. The combined group will undertake progressive treadmill walking speed while performing a cognitive task with rhythmic auditory cueing (i.e., 110% of baseline cadence). The cognitive group will receive cognitive training while walking at a progressive speed on the treadmill. The treadmill-alone group will train only in treadmill walking with progressive speed adjusted weekly. A blinded assessor will administer three assessments. All participants will be examined for gait and cognitive performance under single-task (walking only, Stroop task only) and dual-task conditions (walking while performing the Stroop task) at baseline, post-intervention, and one-month follow-up. The primary outcome measures are gait and cognition under single- and dual-task conditions. The secondary outcome measures are the 6-minute Walk Test, Mini-BESTest, Stroke Impact Scale, and Walking Ability Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with first-time stroke;
* more than 6 months after stroke onset;
* able to walk 10 meters;
* no severe vision, hearing, or speech impairments;
* understand and follow the instructions and sign the Informed Consent Form;
* older than 20 years old.

Exclusion Criteria:

* orthopedic problems affecting walking or other diseases that may interfere with study participation;
* a score of less than 24 on the mini-mental state examination (MMSE);
* severe balance disorder with a total score of less than 45 points Berg Balance Scale.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
walking speed (m/s) under single-task walking and dual-task walking with the Stroop task | baseline, after 4-week intervention, one-month follow-up
  Participants will walk 10 meters at their preferred speed with and without the Stroop task twice, respectively. The spatiotemporal gait parameters will be examined using Physilog® sensors (Gait Up, Switzerland) and analyzed by the Gait Analysis Package software on the USB key. Walking speed (m/s) is the mean speed of forward walking, calculated in meters per second.
swing phase asymmetry under single-task walking and dual-task walking with the Stroop task | baseline, after 4-week intervention, one-month follow-up
  Swing phase asymmetry (%) is the ratio of swing which compares the time in the air for the two feet, in percent.
stride length asymmetry under single-task walking and dual-task walking with the Stroop task | baseline, after 4-week intervention, one-month follow-up
  Stride length asymmetry (%) is the ratio of stride length which compares the stride length for the two feet, in percent. A perfect symmetry outputs a value of 0%.
cognitive composite score | baseline, after 4-week intervention, one-month follow-up
  The Stroop task is the commonly utilized dual-task paradigm and measures executive function and response inhibition, which plays a vital role during walking. Therefore, the Stroop task will be selected to assess cognitive dual-task walking. The Stroop task will be performed while sitting and walking to assess executive function under single-task and dual-task conditions. The following is the formula for calculating the cognitive composite score: Cognitive composite score of the Stroop task = [Accuracy(%)/Reaction time(milliseconds)] * 100. The better the cognitive performance of the Stroop task, the higher the cognitive composite score.
  The instructions for the dual-task walking (walking + Stroop) are designed to encourage neutral prioritization between the two tasks ("walk at the preferred speed while performing the Stroop task as accurately and quickly as you can").

SECONDARY OUTCOMES:
Task-specific dual-task interference | baseline, after 4-week intervention, one-month follow-up
  Task-specific dual-task interference is calculating the motor (i.e., walking speed) or cognitive dual-task effect (DTE), which relates dual-task performance to single-task performance. For assessing dual-task interference, quantifies the combined interference of the motor and the cognitive tasks may be a more comprehensive measure of dual-task effect to provide a more accurate picture of gait automaticity
Automaticity | baseline, after 4-week intervention, one-month follow-up
  Automaticity is based on the combined interference of both motor (i.e., walking speed) and cognitive DTE. The combined dual-task effect (cDTE) is a measure that quantifies automaticity while performing a dual-task.
6-minute Walking test, 6MWT | baseline, after 4-week intervention, one-month follow-up
  The 6MWT is used to measure participants' walking capacity and walking endurance.The participants are asked to walk for six minutes at their own pace, resting or slowing down as needed, and the total distance (meters) of walking in six minutes.
Stroke impact scale, SIS | baseline, after 4-week intervention, one-month follow-up
  The SIS was developed to measure the quality of life after a stroke. The SIS 3.0 has eight domains: strength, hand function, mobility, activities of daily living/instrumental activities of daily living (i.e., ADLs and IADLs), memory and thinking, communication, emotion, and social participation. Scores for each domain range from 0 to 100, and higher scores indicate a better health-related quality of life. Lower scores indicate more incredible difficulty in task completion during the past week or past two weeks, or past four weeks. Eight items on the social participation domain and eight items on the mobility domain of the SIS will be used to measure the social participation of individuals with chronic stroke in this study.
Mini-Balance Evaluation System Test, Mini-BESTest | baseline, after 4-week intervention, one-month follow-up
  The Mini-BESTest is a reliable and valid tool for evaluating balance in people with chronic stroke. It consists of 14 items and includes four subscales: anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait. Each test item is rated on a three-point ordinal scale (0-2, 0=severe, 1=moderate, and 2=normal), with the total score ranging between 0 and 28 points.
Walking ability questionnaire | baseline, after 4-week intervention, one-month follow-up
  Walking ability questionnaire was designed to provide a more detailed assessment of the individual's social limitations due to reduced walking ability. The questionnaire will be administered by a research assistant to rate the participant's current customary mobility of 19 ambulatory activities performed in the home (8 items) and community (11 items). Each item of walking ability is rated on a five-point ordinal scale (0-4, 0=unable to walk, 1=depend on wheel chair, 2=need assistance, 3=walking under supervision, and 4=independent walking), with the total score ranging between 0 and 76 points.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ling Chuang, Ph.D., Principal Investigator — Chang Gung University
Locations (1):
- Mackay Memory Hospital, Taipei, Taiwan